CLINICAL TRIAL: NCT03232268
Title: HLA-mismatched Microtransplantation Without Immunosuppressive Treatment in Patients With Myeloid Hemopathies
Acronym: MICROSTEM
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MICROSTEM- IPC 2016-013
Record Dates: First submitted 2017-07-25; First posted 2017-07-27 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes
Keywords: Microtransplantation; Myeloid Hemopathy
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HLA-mismatched microtransplantation (Experimental): HLA-mismatched microtransplantation without immunosuppressive treatment
  Interventions: Biological: HLA-mismatched microtransplantation

INTERVENTIONS:
Biological: HLA-mismatched microtransplantation — 3 administrations of hematopoietic stem cells without immunosupression

SUMMARY:
This study aims at evaluating the safety of an approach based on HLA-mismatched Microtransplantation without immunosuppressive treatment in patients With myeloid hemopathies who are ineligible to conventional allograft

ELIGIBILITY:
Inclusion Criteria:

* Age> or = 65 years with a myeloid hemopathy in Complete Remission or Complete remission with incomplete hematological recovery or Age<65 years with an ineligibility to allograft (contraindication to conditioning)
* HLA-partially matched family donors
* Affiliated to(or beneficiary of) the Social Security
* Informed consent signed

Exclusion Criteria:

* AML3
* Previous Hematopoietic Stem Cell TRansplantation
* Uncontrolled infection -PS>3 -Other progressive cancer
* Psychiatric disease
* Vulnerable person or unable to provide informed consent
* Emergency
* Unable to comply with required study follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-03-09 (Actual); Primary Completion 2027-03-09 (Estimated); Study Completion 2027-03-09 (Estimated)

PRIMARY OUTCOMES:
Occurrence of acute Graft versus Host disease after a HLA-mismatched transplantation without an immunosuppressive treatment | 100 days after transplantation
  Cumulative incidence of acute GVH (grade 1 to 4)

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Paoli Calmettes, Marseille, Bouches du Rhône, France